CLINICAL TRIAL: NCT03699696
Title: A Pilot Analysis of the Association Between Anesthesia Induction Dosing and Acute Kidney Injury (AKI) in the Elderly Population
Brief Title: A Pilot Analysis of the Association Between Anesthesia Induction Dosing and AKI in the Elderly Population
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000023458
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Acute Kidney Injury; Hypotension; Anesthesia; Adverse Effect
Keywords: acute kidney injury; hypotension; anesthetic dosing; induction; elderly
MeSH Terms: conditions — Acute Kidney Injury; Hypotension | interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 65-75 years of age: Patients who are between the ages of 65 and 75, including 65 but not including 75, and receive propofol for induction of anesthesia.
  Interventions: Drug: Propofol
- 75-85 years of age: Patients who are between the ages of 75 and 85, including 75 but not including 85, and receive propofol for induction of anesthesia.
  Interventions: Drug: Propofol
- 85+ years of age: Patients who are 85 years of age or older, and receive propofol for induction of anesthesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Induction of anesthesia prior to surgery with propofol
  Other Names: Diprivan

SUMMARY:
This study proposes to perform a pilot observational study looking at the doses of propofol used for the induction of general anesthesia and its association with the development of hypotension and AKI among elderly patients at YNHH.

DETAILED DESCRIPTION:
The first stage of this study proposes to perform a pilot observational study looking at the doses of propofol used for the induction of general anesthesia. We will determine the percent (as a function of age, Elixhauser score, ASA status) of patients who receive more than the FDA approved induction dosage. We estimate 30% with the power defined as the width of the 95 percent confidence interval around that number that is given by 80% power and n=500.

In the second stage, the investigators will look at the association between dose and the development of hypotension (in the time after induction and before surgical incision) and post-operative AKI among elderly patients at YNHH while controlling for age, Elixhauser score, and ASA status. The results of this study will also hopefully be used in a quality improvement project to prevent overdosing of the elderly patient population with induction anesthetic.

Hypothesis 1: Elderly patients are being overdosed (per FDA guidelines) with anesthetic agents for induction of general anesthesia.

Hypothesis 2: Overdose of anesthetic agents for induction of general anesthesia in the elderly population leads to an increased chance of developing AKI.

Hypothesis 3: Overdose of anesthetic agents for induction of general anesthesia in the elderly population leads to an increased chance of developing hypotension post-induction, which may contribute to development of AKI or vice-versa.

This research will be done via analysis of data and associated records contained in the Multicenter Perioperative Outcomes Group databases at Yale (the latter is a research database approved under HIC#1206010438).

The possible risks are primarily the risk to privacy that is inherent in any retrospective chart review. The benefit may be to suggest areas for quality improvement in induction practices for elderly patients at YNHH and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 65 or older who underwent induction of general anesthesia at YNHH
* Only first surgery for each patient within the time period is counted
* Only include patients who underwent intubation
* Only include patients who underwent induction by propofol bolus
* Only include patients who got at least 0.3mg/kg of propofol

Exclusion Criteria:

* Patients under the age of 65, patients who underwent monitored anesthetic care/conscious mediation for their procedures.
* Patients with renal failure and/or chronic kidney disease
* Patients who have a pre-operative systolic blood pressure <100

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients who underwent induction of general anesthesia at YNHH, looking specifically at elderly patients undergoing gynecology-oncology surgeries with intubation and propofol induction.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
Overdose | Between time of induction of anesthesia and surgical incision as detailed in the patient's anesthesia record
  Percentage of patients >=65 who received greater than the FDA approved induction dosage of propofol

SECONDARY OUTCOMES:
Hypotension | Between time of induction of anesthesia and surgical incision as detailed in the patient's anesthesia record
  Mean arterial pressure of less than 60mmHg
Acute kidney injury | Within 7 days postoperatively
  AKI identifies when there is an increase of 1.5 times the baseline serum creatinine observed in first 7 postoperative days OR when the baseline creatinine increases greater than or equal to 0.3 mg/dl in 48 hours after anesthesia end. Baseline serum creatinine is defined as the most recent serum creatinine resulted in the last 60 days preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Y Chen, BS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen EY, Michel G, Zhou B, Dai F, Akhtar S, Schonberger RB. An Analysis of Anesthesia Induction Dosing in Female Older Adults. Drugs Aging. 2020 Jun;37(6):435-446. doi: 10.1007/s40266-020-00760-3. PMID 32300966